CLINICAL TRIAL: NCT01517152
Title: Spanish Translation and Linguistic Validation of the Patient- Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Brief Title: Testing a Spanish Version of a Patient Toxicity Questionnaire
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912040; 12-C-N040
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-10-09

CONDITIONS: Breast Cancer; Colon Cancer; Lung Cancer; Lymphoma; Myeloma
Keywords: Symptoms; Patient-Reported Outcomes; Linguistic Validation; Toxicity; PRO-CTCAE; Adverse Events; Translation; Questionnaire
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* The Common Terminology Criteria for Adverse Events (CTCAE) is a list of toxicities and side effects that may occur when people are having cancer treatment. Doctors and nurses use this list to describe the side effects patients experience from cancer treatment. We have developed a questionnaire to ask people having cancer treatment directly about common symptoms and side effects and to supply this information to their doctors and nurses. This questionnaire is known as PRO-CTCAE and is completed by a patient.
* PRO-CTCAE was originally developed in English. Researchers want to develop a Spanish version of the patient questionnaire. To test whether the questions are well understood and whether it is easy to complete the questionnaire, the researchers will interview individuals whose primary language is Spanish and who are being treated for different types of cancer.

Objectives:

- To test a Spanish version of the PRO-CTCAE questionnaire.

Eligibility:

- Latinos at least 18 years of age who are having or have recently finished cancer treatments and whose main language is Spanish

Design:

* Participants will complete a questionnaire in Spanish with selected questions from the translated PRO-CTCAE. They will discuss their answers and any difficulties they might have had in understanding or answer the questions with an interviewer, who will take notes and record comments and suggestions.
* Literacy is not required for this study. Participants may opt to have the questions read aloud to them by an interviewer.

DETAILED DESCRIPTION:
This study describes a study to assess a newly created Spanish version of the National Cancer Institute s (NCI s) patient toxicity questionnaire, the Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), via semi-structured interviews among Spanish-speaking patients with cancer in the United States.

Background:

The NCI s PRO-CTCAE initiative has developed and preliminarily validated a library of items in English intended for patient self-reporting of treatment toxicity and symptoms during participation in cancer clinical trials. These items have also been translated into Spanish, using a methodology consistent with internationally agreed-upon guidelines for developing global translations.

Objective:

To linguistically validate a Spanish-language version of PRO-CTCAE symptom items to assure that they are culturally, semantically, and linguistically proficient to the native Spanish-speaking population with cancer in the United States.

Eligibility:

Research participants must be (i) 18 years or older; (ii) able to provide informed consent; (iii) currently undergoing systemic cancer treatment or immediately post-treatment; (iv) speak Spanish as their primary language.

Design:

Two rounds of PRO-CTCAE questionnaire administration followed by cognitive interviews will be conducted with Spanish speakers residing in the US. Between 40-60 interviews will be conducted in the first round, and up to 20 additional interviews will be conducted in an optional second round; total accrual will be 80 participants. Participating sites have been selected to assure access to participants from a range of Spanish-speaking countries of origin, and those with lower levels of educational attainment and acculturation.

Cognitive interviewing methodology provides an approach to determining that language adaptations produced through forward and back translation are conceptually equivalent to the English source document, and cross-culturally valid. Data derived from cognitive interviewing permit a conclusion that item meanings are qualitatively equivalent after translation and across individuals, and permit refinement, as necessary, to render terminologies and phrasing that are culturally acceptable and relevant to the target population.

A large number of PRO-CTCAE symptom items will be evaluated in this study, and in addition, several of the items are gender-specific. To minimize patient burden and ensure that the item pool is uniformly evaluated relative to participant gender, education, acculturation and country of origin, items have been distributed across four questionnaires, each matched with a tailored interview schedule. Each participant will complete one questionnaire and participate in one interview.

Interviewers are Bachelor- and Masters-prepared research staff who are bilingual and have experience with cognitive interviewing in clinical research and/or cancer treatment settings.

Interview summaries will be produced in English by each interviewer; audiotapes will be reviewed as necessary. These summaries together with relevant field notes will be assembled into a report, and used to further refine the translated PRO-CTCAE items.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be 18 years or older and be able to provide informed consent.
* Participants must be patients being followed for clinical care at one of the collaborating sites, and must be either currently undergoing or having completed treatment for cancer in the previous 6 months.
* Participants must be native Spanish-speakers.
* Participants must be able either to read and understand the items in Spanish or to hear and understand and respond to the items when read to them verbatim in Spanish.

EXCLUSION CRITERIA:

* Cognitive impairment as determined by the patient s Physician or Nurse which renders them unable to understand the items or report on his/her symptoms from the last 7 days.
* If participants request to have the consent form in English, they will not be eligible for participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-01-04; Study Completion 2018-10-09

PRIMARY OUTCOMES:
Perceptions of the clarity and ease of response to a series of questions | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Mitchell, C.R.N.P., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Basch E. The missing voice of patients in drug-safety reporting. N Engl J Med. 2010 Mar 11;362(10):865-9. doi: 10.1056/NEJMp0911494. No abstract available. PMID 20220181
- [Background] Bonomi AE, Cella DF, Hahn EA, Bjordal K, Sperner-Unterweger B, Gangeri L, Bergman B, Willems-Groot J, Hanquet P, Zittoun R. Multilingual translation of the Functional Assessment of Cancer Therapy (FACT) quality of life measurement system. Qual Life Res. 1996 Jun;5(3):309-20. doi: 10.1007/BF00433915. PMID 8763799
- [Background] Johnson TP. Methods and frameworks for crosscultural measurement. Med Care. 2006 Nov;44(11 Suppl 3):S17-20. doi: 10.1097/01.mlr.0000245424.16482.f1. PMID 17060823